CLINICAL TRIAL: NCT00894361
Title: A Randomized Prospective Comparison of Mobile-Bearing and Fixed-Bearing (All-Polyethylene Tibia) Cruciate-Substituting Total Knee Arthroplasty (TKA) Designs
Brief Title: Comparison of Mobile-Bearing and Fixed-Bearing All-Polyethylene Tibia Total Knee Designs
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI/study coordinator retired due to personal family health matters; study sponsor withdrew funding. Study terminated and no data collected or analyzed
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Depuy, Inc. (Industry)
Responsible Party: Principal Investigator, Terence J. Gioe, M.D., Chief, Dept. of Orthopaedic Surgery, Minneapolis VAMC, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MVA-3028
Record Dates: First submitted 2009-03-24; First posted 2009-05-07 (Estimated); Results first posted 2009-05-07 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Osteoarthritis, Knee
Keywords: knee arthritis; total knee arthroplasty; total knee replacement; mobile bearing design; all-polyethylene tibia
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rotating-platform design TKA (Active Comparator): patients who were randomized to receive the rotating platform mobile-bearing TKA design
  Interventions: Procedure: TKA surgery with the rotating platform mobile-bearing knee design
- all-polyethylene tibia design TKA (Active Comparator): patients who were randomized to receive the all-polyethylene tibial component design
  Interventions: Procedure: TKA surgery with the all-polyethylene tibia knee design

INTERVENTIONS:
Procedure: TKA surgery with the rotating platform mobile-bearing knee design — Depuy Sigma RP rotating platform design
  Arms: rotating-platform design TKA
Procedure: TKA surgery with the all-polyethylene tibia knee design — Depuy Sigma fixed-bearing design with all-polyethylene tibia
  Arms: all-polyethylene tibia design TKA

SUMMARY:
This study will be designed to compare prospectively, in a randomized fashion, the clinical, functional, and radiographic results of a nonmodular (all-polyethylene tibi/AP) fixed-bearing posterior cruciate substituting design with a modular posterior cruciate substituting rotating platform (RP) design for total knee arthroplasty. Comparing these two designs will afford the investigators information in the following areas:

1. Does a RP design offer improvement in range of motion over a AP design?
2. Does a RP design have improved wear characteristics over a nonmodular AP design?
3. Is there a clear clinical advantage to the RP design that justifies its increased cost?

Answering these questions will allow surgeons to use RP designs appropriately in different demand populations.

This study was designed to address the questions of whether an RP design offers improvement in ROM, Knee Society scores, Western Ontario and McMaster Universities Index of Osteoarthritis (WOMAC) scores, selected Medical Outcomes Short-Form Health Survey Short Form-36 (SF-36) scores or radiographic measures, over an APT design. The investigators' primary hypothesis was that there would be no difference in these outcome measures at a minimum two year followup. A secondary hypothesis based on the anticipated long-term followup of this group was that there would be no difference in implant survival.

ELIGIBILITY:
Inclusion Criteria:

* generally accepted clinical and radiographic criteria for primary total knee arthroplasty

Exclusion Criteria:

* substantial angular deformity or bony deformity requiring structural grafting or modular augmentation were excluded at the discretion of the principle investigator
* patients whose mental function precluded them from responding to our standard questionnaires

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2001-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence J Gioe, M.D., Principal Investigator — Minneapolis VAMC, Dept. of Orthopaedic Surgery
Locations (1):
- Minneapolis VAMC, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Gioe TJ, Glynn J, Sembrano J, Suthers K, Santos ER, Singh J. Mobile and fixed-bearing (all-polyethylene tibial component) total knee arthroplasty designs. A prospective randomized trial. J Bone Joint Surg Am. 2009 Sep;91(9):2104-12. doi: 10.2106/JBJS.H.01442. PMID 19723986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: October 1, 2001 to January 1, 2007 recruitment period from the Minneapolis VAMC Orthopaedic Clinic
Pre-assignment Details: Patients that were recruited but not enrolled either failed the inclusion criteria or elected not to participate
Groups:
- Rotating-platform Design Total Knee Arthroplasty (TKA): patients who were randomized to receive the rotating platform mobile-bearing TKA design
- All-polyethylene Tibia Design Total Knee Arthroplasty (TKA): patients who were randomized to receive the all-polyethylene tibial component design
Period: Overall Study
Arm/Group | Rotating-platform Design Total Knee Arthroplasty (TKA) | All-polyethylene Tibia Design Total Knee Arthroplasty (TKA)
Started | 200 | 200
Completed | 176 | 136
Not Completed | 24 | 64
Not completed — deaths and less than 2 years followup | 24 | 64

BASELINE CHARACTERISTICS:
Groups:
- Rotating-platform Design Total Knee Arthroplasty (TKA): patients who were randomized to receive the rotating platform mobile-bearing total knee arthroplasty (TKA) design
- Total: Total of all reporting groups
Arm/Group | Rotating-platform Design Total Knee Arthroplasty (TKA) | All-polyethylene Tibia Design Total Knee Arthroplasty (TKA) | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 79 | 74 | 153
  >=65 years | 121 | 126 | 247
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 195 | 193 | 388
Region of Enrollment [Number; unit: participants]
  United States | 200 | 200 | 400
range of motion of knee [Mean (Standard Deviation); unit: degrees] | 113.7 (1.0) | 111.9 (1.1) | 112.8 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Knee Postoperative Range of Motion (ROM) at 2 Years
Description: range of motion of the knee postoperatively at 2 years
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rotating-platform Design Total Knee Arthroplasty (TKA) | All-polyethylene Tibia Design Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 176 | 136
degrees | 110.4 (0.8) | 111.9 (0.9)

2. Secondary Outcome: Survival of the Implants to Subject Death or Implant Removal
Time Frame: 10 or more years
Population: PI/study coordinator retired due to personal family health matters and study sponsor withdrew funding. Study was terminated and no data was collected or analyzed from any participant for this outcome measure.
Arm/Group | Rotating-platform Design TKA | All-polyethylene Tibia Design TKA
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 Years
Description: PI/study coordinator retired due to personal family health matters and study sponsor then withdrew funding. Study terminated and no data was collected or analyzed from any participant.
Arm/Group | Rotating-platform Design Total Knee Arthroplasty (TKA) | All-polyethylene Tibia Design Total Knee Arthroplasty (TKA)
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/200
Other Adverse Events (participants affected / at risk) | 0/200 | 0/200

LIMITATIONS AND CAVEATS:
PI/study coordinator retired due to personal family health matters and study sponsor then withdrew funding. Study terminated and no data was collected or analyzed from any participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No